CLINICAL TRIAL: NCT02763267
Title: Study of Pregnancy Regulation of Insulin and Glucose
Acronym: SPRING
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Camille Elise Powe,M.D., Co-Director, MGH Diabetes in Pregnancy Program, Massachusetts General Hospital
Other Study IDs: 2015P002447
Record Dates: First submitted 2016-02-17; First posted 2016-05-05 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Insulin sensitivity; Insulin secretion; Pregnancy; Placental proteins
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, DNA, plasma, serum. With subject consent: maternal cord blood, urine, DNA, fetal cord blood, neonatal DNA, placental tissue, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant Women: Pregnant women with history of GDM or at risk for diabetes mellitus will enter study during first trimester (4-14 weeks) and receive an oral glucose tolerance test (OGTT) at baseline, mid-pregnancy, and at delivery.
  Interventions: Other: Oral glucose tolerance test
- Nonpregnant Women: Nonpregnant women with a history of GDM will undergo an OGTT at baseline.
  Interventions: Other: Oral glucose tolerance test

INTERVENTIONS:
Other: Oral glucose tolerance test — 75 gram oral glucose tolerance test (fasting) at: Visit 1 (pregnant [4-14 weeks gestation] and nonpregnant women); Visit 2 (pregnant subjects only at 24-28 weeks gestation); Visit 3 (pregnant subjects only at 6-12 weeks postpartum)
  Other Names: OGTT

SUMMARY:
It is unknown whether beta cell dysfunction and insulin resistance in Gestational Diabetes Mellitus (GDM) is representative of a chronic maternal defect, unmasked by pregnancy, or whether it is the result of an imbalance of a placental hormones. Undiscovered placental factors which vary between pregnancies likely contribute to the pathogenesis of GDM. To elucidate the pathophysiology underlying GDM, the investigators will attempt to discover these factors and characterize pregnancy-associated changes in insulin secretion and sensitivity in women with and without GDM.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) complicates 3-7% of pregnancies in the United States and is associated with perinatal morbidity and a high risk of future maternal type 2 diabetes. Current prevention and treatment of GDM relies on techniques developed in the type 2 diabetes population, without regard to unique physiology in pregnancy. GDM occurs in the setting of profound pregnancy changes in glucose metabolism: late pregnancy is normally characterized by marked insulin resistance. In order to maintain normal glucose levels and avoid GDM, pancreatic beta cells must augment insulin secretion to compensate. Women with GDM have inadequate beta-cell compensation for pregnancy-induced insulin resistance, resulting in hyperglycemia. It is unknown whether beta cell dysfunction and insulin resistance in GDM is representative of a chronic maternal defect, unmasked by pregnancy, or whether it is the result of an imbalance of a placental hormones. Undiscovered placental factors which vary between pregnancies likely contribute to the pathogenesis of GDM. Discovery of these factors and elucidation of the pathophysiology underlying GDM will allow for the development better GDM-specific prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Women, age 18-44, non-pregnant OR in the 1st trimester of pregnancy (4-14 weeks gestation),
* Who had GDM in a previous pregnancy
* At risk for diabetes mellitus, as specified by the American Diabetes Association (ADA):
* BMI ≥ 25 kg/m2 (or BMI ≥ 23 kg/m2 if Asian-American) PLUS one or more of the following:

  * history of giving birth to a neonate weighing > 9 lbs
  * first-degree family member with diabetes mellitus
  * high-risk ethnic or racial group (African-American, Hispanic, Native American, Asian-American, or Pacific Islander)
  * polycystic ovary syndrome
  * hypertension, dyslipidemia if known (HDL<45 and/or triglyceride level >250), or cardiovascular disease
  * physical inactivity

Exclusion Criteria:

* Known pre-existing diabetes mellitus, based on patient report or medical record review
* A1C ≥ 6.5%, detected at study visit 1
* Use of medications known to affect glucose tolerance including corticosteroids, metformin, sulfonylureas, and others as determined by the investigators.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 150 Pregnant Women with history of GDM or at risk for diabetes mellitus and 200 Nonpregnant Women with history of GDM
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Insulin secretory response | 1st trimester (gestational weeks 4-14)
  Insulin secretory response to a glucose load (insulinogenic index), adjusted for differences in insulin resistance, in pregnant women in the 1st trimester will be compared to the insulin secretory response in non-pregnant women

SECONDARY OUTCOMES:
Insulin secretory response | Mid-pregnancy (gestational weeks 24-28)
  Insulin secretory response to a glucose load (insulinogenic index), adjusted for differences in insulin resistance, in pregnant women at 24-28 weeks gestation will be compared to the insulin secretory response in non-pregnant women
Change in insulin secretory response | 1st trimester to 24-28 weeks gestation
  Change in insulin secretory response to a glucose load (insulinogenic index) between 1st trimester and 24 to 28 weeks gestation, adjusted for changes in insulin resistance, in pregnant women who do and do not develop GDM
Change in insulin secretory response | 1st trimester to postpartum (up to 12 weeks post-partum or up to 50 weeks after the first trimester visit, whichever comes first)
  Change in insulin secretory response to a glucose load (insulinogenic index) between 1st trimester and postpartum, adjusted for changes in insulin resistance, in pregnant women who do and do not develop GDM

CONTACTS AND LOCATIONS:
Overall Officials: Ravi I Thadhani, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rosenberg EA, Seely EW, James K, Soffer MD, Nelson S, Nicklas JM, Powe CE. Carbohydrate Intake and Oral Glucose Tolerance Test Results in the Postpartum Period. J Clin Endocrinol Metab. 2023 Sep 18;108(10):e1007-e1012. doi: 10.1210/clinem/dgad234. PMID 37097924